CLINICAL TRIAL: NCT00436111
Title: Characterization of Macroprolactinemia
Status: Completed | Type: Observational
Sponsor: Kansai Medical University (Other)
Other Study IDs: KK-2007-1
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Last update posted 2007-02-16 (Estimated); Status verified 2007-02

CONDITIONS: Hyperprolactinemia
Keywords: hyperprolactinemia; autoantibody
MeSH Terms: conditions — Hyperprolactinemia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to clarify the nature of macroprolactin which has recently been highlighted because of the high prevalence and a diagnostic pitfall of hyperprolactinemia. The results of this study are beneficial for the patients to whom unnecessary medications and unnecessary radiological examinations have been performed.

We used the remained serum samples taken for routine prolactin determination during the past several years. Since the blood was basically taken to examine the causes of hyperprolactinemia and only remained serum samples were used for this study, the Ethics Committee of Kobe City General Hospital judged that it was not required to obtain approval number.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hyperprolactinemia

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-01; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Hattori, M.D., Ph.D., Study Chair — Department of Pharmacology, Kansai Medical University
Locations (1):
- Kansai Medical University, Osaka, Osaka, Japan

REFERENCES:
- [Result] Hattori N, Nakayama Y, Kitagawa K, Ishihara T, Saiki Y, Inagaki C. Anti-prolactin (PRL) autoantibody-binding sites (epitopes) on PRL molecule in macroprolactinemia. J Endocrinol. 2006 Aug;190(2):287-93. doi: 10.1677/joe.1.06871. PMID 16899562
- [Result] Hattori N, Ikekubo K, Nakaya Y, Kitagawa K, Inagaki C. Immunoglobulin G subclasses and prolactin (PRL) isoforms in macroprolactinemia due to anti-PRL autoantibodies. J Clin Endocrinol Metab. 2005 May;90(5):3036-44. doi: 10.1210/jc.2004-1600. Epub 2005 Feb 1. PMID 15687336
- [Result] Hattori N, Inagaki C. Anti-prolactin (PRL) autoantibodies cause asymptomatic hyperprolactinemia: bioassay and clearance studies of PRL-immunoglobulin G complex. J Clin Endocrinol Metab. 1997 Sep;82(9):3107-10. doi: 10.1210/jcem.82.9.4250. PMID 9284753
- [Result] Hattori N, Ishihara T, Ikekubo K, Moridera K, Hino M, Kurahachi H. Autoantibody to human prolactin in patients with idiopathic hyperprolactinemia. J Clin Endocrinol Metab. 1992 Nov;75(5):1226-9. doi: 10.1210/jcem.75.5.1430082.